CLINICAL TRIAL: NCT00684502
Title: A Phase I, Single-centre, Randomised, Double-blind, Parallel Group, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD2066 in Young and Elderly Healthy Subjects After Oral Multiple Ascending Doses
Brief Title: Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD2066 in Young and Elderly Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Rolf Karlsten, M.D., Medical Science Director, Emerging Neuroscience, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D0475C00002; EudractCT 2007-005524-33
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2008-12

CONDITIONS: Pain
Keywords: Safety; tolerability; AZD2066; Pain conditions
MeSH Terms: conditions — Pain | interventions — AZD2066

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Oral solution.
  Interventions: Drug: AZD2066
- 2 (Placebo Comparator): Oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2066 — Oral solution administered orally once per day on day 1, and then day 3 through to day 12. Specific dose depends on dose panel.
  Arms: 1
Drug: Placebo — Administered orally as a solution once per day on day 1, and then day 3 through to day 12.
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of AZD2066 using multiple escalating dose panels. There will be separate panels for young healthy volunteers and elderly healthy volunteers. Each panel will contain 10 volunteers who will randomly receive AZD2066 or placebo. One panel will be run at a time with a fixed dose given. After the completion of each panel, a Safety Review Committee will decide if the study can proceed to the next dose panel.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent
* Clinically normal physical findings and laboratory values as judged by the investigator and a normal resting ECG.

Exclusion Criteria:

* History of somatic disease/condition, which may interfere with the objectives of the study, as judged by the investigator.
* History of previous or ongoing psychiatric disease/condition including psychosis, affective disorder, anxiety disorder, borderline state and personality disorder.
* Intake of medicine (except occasional paracetamol or nasal spray) within first 2 weeks before first administration of study drug.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AZD2066 by assessment of vital signs, laboratory variables and ECG | Assessments taken at visit 1 (enrolment), defined time points pre dose and post dose during visit 2 (residential period): days -1 through to day 15 and follow up visit 3

SECONDARY OUTCOMES:
Safety and tolerability of AZD2066 by assessment of adverse events | Non serious adverse events will be collected from the start of Visit 2 until the end of the study. Serious adverse events will be collected from signing of consent until end of study.
Investigate PK profile (including dose proportionality, degree of accumulation and time dependancy) of AZD2066 (and possible relevant metabolites). | PK sampling taken at defined timepoints during residential period and follow-up.
Investigate CNS effects of AZD2066 | Psychometric test battery performed at defined timepoints during the residential period. Test on day -1 for training purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Fransson, MD, Principal Investigator — AstraZeneca R&D SödertäljeMedical Science, CPU C2:84Karolinska University Hospital HuddingeSE-141 86 Stockholm, Sweden; Lars Stahle, MD, PhD, Study Chair — AstraZeneca R&D Södertälje Medical Science S-151 85 Södertälje Sweden
Locations (1):
- Research Site, Stockholm, Sweden